CLINICAL TRIAL: NCT04966741
Title: A Phase 3 Multi-Center, 1-Year, Open-Label Study of Setmelanotide in Pediatric Patients Aged 2 to <6 Years of Age With Rare Genetic Causes of Obesity
Brief Title: Setmelanotide in Pediatric Participants With Rare Genetic Diseases of Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-033
Record Dates: First submitted 2021-03-29; First posted 2021-07-19 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Bardet-Biedl Syndrome; POMC Deficiency Obesity; PCSK1 Deficiency Obesity; LEPR Deficiency Obesity
Keywords: Bardet Biedl Syndrome; POMC Deficiency; PCSK1; LEPR; Obesity; Pediatric Obesity
MeSH Terms: conditions — Bardet-Biedl Syndrome; Proopiomelanocortin Deficiency; Obesity; Pediatric Obesity | interventions — setmelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Setmelanotide: PPL Group (Experimental): Participants with POMC)/PCSK1/LEPR biallelic mutations collectively referred to as PPL received setmelanotide at a dose of 0.5 milligrams (mg) per day (QD) via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label long-term extension (LTE) trial with setmelanotide.
  Interventions: Drug: Setmelanotide
- Setmelanotide: BBS Group (Experimental): Participants with BBS received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label long-term extension (LTE) trial with setmelanotide.
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — SC injection once daily.
  Other Names: IMCIVREE

SUMMARY:
This is a phase 3 open-label, clinical study to evaluate the efficacy, safety and tolerability of setmelanotide over 1 year of treatment, in pediatric participants aged 2 to <6 years with obesity due to either biallelic variants of the pro-opiomelanocortin (POMC), proprotein convertase subtilisin/kexin type 1 (PCSK1) or leptin receptor (LEPR) genes or Bardet-Biedl Syndrome (BBS).

DETAILED DESCRIPTION:
Pediatric participants aged 2 to <6 years with obesity due to either biallelic variants of the POMC, PCSK1 or LEPR genes or BBS will be enrolled into this phase 3 open-label clinical trial at one of approximately 8 clinical centers in North America, Europe, or Australia. All participants will be assigned to receive setmelanotide via daily subcutaneous (SC) injection for 1 year.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have obesity due to either:

   1. POMC, PCSK1, or LEPR deficiency, confirmed by genetic testing demonstrating biallelic variants that are interpreted as pathogenic, likely pathogenic, or of undetermined significance (VUS) by the American College of Medical Genetics and Genomics criteria (ACMG), or
   2. BBS confirmed clinical and genetic diagnosis
2. Age between 2 to <6 years at the time of informed consent
3. Obesity, defined as body mass index (BMI) ≥97th percentile for age and gender and body weight of at least 15 kilograms (kg) at the time of enrollment.
4. Symptoms or behaviors of hyperphagia
5. Parent or guardian of study participant is able to understand and comply with the requirements of the study (including QD injection regimen and all other study procedures) and is able to understand and sign the written consent/assent.

Key Exclusion Criteria

1. Glycated hemoglobin (HbA1c) >9.0% at screening
2. History of significant liver disease
3. Glomerular filtration rate (GFR) <60 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2)
4. History or close family history of melanoma, or participant history of oculocutaneous albinism.
5. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion)
6. Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
7. Previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide.
8. Significant hypersensitivity to any excipient in the study drug.
9. Inadequate hepatic function
10. Any other uncontrolled endocrine, metabolic or medical condition(s) known to impact body weight

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (6):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Columbia University Medical Center, Division of Pediatric Endocrinology, Diabetes and Metabolism, New York, New York
  - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Sydney Children's Hospital, Randwick, Australia
- Hospital Infantil Niño Jesus, Madrid, Spain
- Addenbrooke's Hospital, Wellcome Trust-MRC Institute of Metabolic Science, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Argente J, Verge CF, Okorie U, Fennoy I, Kelsey MM, Cokkinias C, Scimia C, Lee HM, Farooqi IS. Setmelanotide in patients aged 2-5 years with rare MC4R pathway-associated obesity (VENTURE): a 1 year, open-label, multicenter, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Jan;13(1):29-37. doi: 10.1016/S2213-8587(24)00273-0. Epub 2024 Nov 13. PMID 39549719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 13 participants screened, 12 participants were enrolled in the study.
Groups:
- Setmelanotide: PPL Group: Participants with pro-opiomelanocortin (POMC)/proprotein convertase subtilisin/kexin type 1 (PCSK1)/leptin receptor (LEPR) biallelic mutations collectively referred to as PPL received setmelanotide at a dose of 0.5 milligrams (mg) per day (QD) via subcutaneous (SC) injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label long-term extension (LTE) trial with setmelanotide.
- Setmelanotide: BBS Group: Participants with Bardet-Biedl syndrome (BBS) received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label LTE trial with setmelanotide.
Period: Overall Study
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Started | 7 | 5
Completed | 6 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Setmelanotide: PPL Group: Participants with POMC/PCSK1/LEPR biallelic mutations collectively referred to as PPL received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label long-term extension (LTE) trial with setmelanotide.
- Setmelanotide: BBS Group: Participants with BBS received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label LTE trial with setmelanotide.
- Total: Total of all reporting groups
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (0.53) | 3.8 (1.30) | 3.6 (0.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 1 | 1
  Race: White | 3 | 4 | 7
  Race: Other | 2 | 0 | 2
  Race: Unknown or Not Reported | 2 | 0 | 2
Body Mass Index (BMI) Z-score [Mean (Standard Deviation); unit: z-score] — BMI Z-scores were based on the World Health Organization's Child Growth Standards 2007. The BMI Z-score indicated the number of standard deviations away from the mean. A Z-score of 0 was equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score (< 0) indicated a reduction in BMI from Baseline whereas an increase of BMI-Z score (> 0) indicated an increase in BMI from Baseline.
  z-score | 10.749 (3.8400) | 4.233 (1.0742) | 8.034 (4.4408)
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kilograms/ square meter (kg/m^2).
  kg/m^2 | 34.347 (7.0673) | 23.716 (3.5184) | 29.918 (7.8559)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 0.2 Reduction of BMI Z-Score From Baseline to Week 52
Description: A "responder" was defined as a decrease from baseline to 52 weeks in the participant's BMI z-score of ≥0.2. BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. The BMI Z-scores were based on the World Health Organization's Child Growth Standards 2007 and indicated the number of standard deviations away from the mean. A Z-score of 0 was equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score (< 0) indicated a reduction in BMI from Baseline whereas an increase of BMI-Z score (> 0) indicated an increase in BMI from Baseline. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline up to Week 52
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Setmelanotide: PPL Group: Participants with POMC/PCSK1/LEPR biallelic mutations collectively referred to as PPL received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight.
- Setmelanotide: BBS Group: Participants with BBS received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight.
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 7 | 5
percentage of participants | 85.7 [54.1 to 100] | 80.0 [28.4 to 99.5]

2. Primary Outcome: Mean Percent Change From Baseline in BMI
Description: Mean percent change from baseline to Week 52 in BMI was reported. BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 6 | 5
percent change | -25.597 (11.4911) | -9.719 (8.8383)

3. Secondary Outcome: Mean Absolute Change From Baseline in BMI Z-score
Description: Mean absolute change from baseline to Week 52 in BMI Z-score was reported. BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. The BMI Z-scores were based on the World Health Organization's Child Growth Standards 2007 and indicated the number of standard deviations away from the mean. A Z-score of 0 was equal to the mean of a reference population (i.e., healthy, age and sex-matched individuals). A decrease of BMI Z-score (< 0) indicated a reduction in BMI from Baseline whereas an increase of BMI-Z score (> 0) indicated an increase in BMI from Baseline. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 6 | 5
Z-score | -5.185 (1.8585) | -1.331 (1.2295)

4. Secondary Outcome: Mean Change From Baseline in Percent of the 95th Percentile of BMI
Description: Mean change from baseline to Week 52 in percent of the 95th percentile of BMI was reported. BMI was calculated using participant's weight and height assessments, using the following formula: BMI = kg/m^2. BMI Percentile-scores are measures of relative weight adjusted for child age and gender. The percent of the BMI 95th percentile score expresses the participant's BMI as a percentage of the Centers for Disease Control (CDC) 95th percentile reference population. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage relative to 95th percentile
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 6 | 5
percentage relative to 95th percentile | -47.595 (17.3280) | -14.462 (13.8571)

5. Secondary Outcome: Mean Change From Baseline in Bone Age
Description: Mean change from baseline to Week 52 in bone age was reported. A standard bone age measurement (of the hand/wrist area) was obtained at the beginning and the end of the trial to monitor for growth related safety concerns. Baseline was defined as the most recent measurement prior to the first administration of study drug.
Time Frame: Baseline, Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 5 | 5
years | 1.020 (1.0733) | 0.700 (0.8367)

6. Secondary Outcome: Number of Participants With Shift From Baseline in Ages & Stages Questionnaires, Third Edition (ASQ-3)
Description: ASQ-3: developmental screening questionnaire that consists of 5 areas: communication, gross motor, fine motor, problem solving, and personal-social. Each area has 6 questions scored as Yes=10 points, Sometimes=5 points, and Not yet=0 points. A child can score between 0-60 points for each area with total score range: 0 to 300; higher scores are indicative of improvement. Total area score is then compared to age-adjusted standardized score cutoff (determined by developers of tool) which indicate whether child's development appears to be on schedule according to these categories: Below=Total analysis score (TAS) is below cutoff. Further assessment with professional may be needed; Monitor=TAS is close to cutoff. Provide learning activities and monitor; Above= TAS is above cutoff, and child's development appears to be on schedule. Shift from baseline for each developmental area of assessment according to these 3 outcome categories was reported. Total score was not applicable.
Time Frame: From Baseline to Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 6 | 5
Participants
  Communication: Baseline (Above): Week 52 (Above) | 5 | 2
  Communication: Baseline (Above): Week 52 (Monitor) | 0 | 0
  Communication: Baseline (Above): Week 52 (Below) | 0 | 0
  Communication: Baseline (Monitor): Week 52 (Above) | 0 | 0
  Communication: Baseline (Monitor): Week 52 (Monitor) | 0 | 1
  Communication: Baseline (Monitor): Week 52 (Below) | 0 | 0
  Communication: Baseline (Below): Week 52 (Above) | 0 | 0
  Communication: Baseline (Below): Week 52 (Monitor) | 0 | 0
  Communication: Baseline (Below): Week 52 (Below) | 1 | 2
  Fine Motor: Baseline (Above): Week 52 (Above) | 4 | 2
  Fine Motor: Baseline (Above): Week 52 (Monitor) | 0 | 0
  Fine Motor: Baseline (Above): Week 52 (Below) | 0 | 0
  Fine Motor: Baseline (Monitor): Week 52 (Above) | 0 | 1
  Fine Motor: Baseline (Monitor): Week 52 (Monitor) | 0 | 0
  Fine Motor: Baseline (Monitor): Week 52 (Below) | 1 | 1
  Fine Motor: Baseline (Below): Week 52 (Above) | 0 | 0
  Fine Motor: Baseline (Below): Week 52 (Monitor) | 0 | 0
  Fine Motor: Baseline (Below): Week 52 (Below) | 1 | 1
  Gross Motor: Baseline (Above): Week 52 (Above) | 1 | 0
  Gross Motor: Baseline (Above): Week 52 (Monitor) | 0 | 0
  Gross Motor: Baseline (Above): Week 52 (Below) | 0 | 0
  Gross Motor: Baseline (Monitor): Week 52 (Above) | 0 | 0
  Gross Motor: Baseline (Monitor): Week 52 (Monitor) | 0 | 0
  Gross Motor: Baseline (Monitor): Week 52 (Below) | 0 | 0
  Gross Motor: Baseline (Below): Week 52 (Above) | 3 | 1
  Gross Motor: Baseline (Below): Week 52 (Monitor) | 0 | 2
  Gross Motor: Baseline (Below): Week 52 (Below) | 2 | 2
  Personal - Social: Baseline (Above): Week 52 (Above) | 3 | 2
  Personal - Social: Baseline (Above): Week 52 (Monitor) | 0 | 0
  Personal - Social: Baseline (Above): Week 52 (Below) | 0 | 0
  Personal - Social: Baseline (Monitor): Week 52 (Above) | 2 | 0
  Personal - Social: Baseline (Monitor): Week 52 (Monitor) | 0 | 0
  Personal - Social: Baseline (Monitor): Week 52 (Below) | 0 | 0
  Personal - Social: Baseline (Below): Week 52 (Above) | 1 | 1
  Personal - Social: Baseline (Below): Week 52 (Monitor) | 0 | 0
  Personal - Social: Baseline (Below): Week 52 (Below) | 0 | 2
  Problem Solving: Baseline (Above): Week 52 (Above) | 4 | 3
  Problem Solving: Baseline (Above): Week 52 (Monitor) | 0 | 0
  Problem Solving: Baseline (Above): Week 52 (Below) | 0 | 0
  Problem Solving: Baseline (Monitor): Week 52 (Above) | 0 | 0
  Problem Solving: Baseline (Monitor): Week 52 (Monitor) | 0 | 0
  Problem Solving: Baseline (Monitor): Week 52 (Below) | 0 | 0
  Problem Solving: Baseline (Below): Week 52 (Above) | 1 | 0
  Problem Solving: Baseline (Below): Week 52 (Monitor) | 1 | 0
  Problem Solving: Baseline (Below): Week 52 (Below) | 0 | 2

7. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline to Week 52 in body weight was reported.
Time Frame: Baseline, Week 52
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 6 | 5
kilograms | -7.139 (5.0834) | -0.327 (2.9572)

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE was defined as any AE that started or worsened in intensity on or after the date of the first administration of study drug.
Time Frame: From first dose of study drug up to Week 56
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 7 | 5
Participants | 7 | 5

9. Secondary Outcome: Number of Participants With TEAEs Graded by Severity
Description: A TEAE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE was defined as any AE that started or worsened in intensity on or after the date of the first administration of study drug. TEAEs were graded according to Common Terminology Criteria for Adverse Events (CTCAE) criteria. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life Threatening; Grade 5- Death related to AE.
Time Frame: From first dose of study drug up to Week 56
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
Number analyzed (Participants) | 7 | 5
Participants
  Mild | 2 | 5
  Moderate | 5 | 0
  Severe | 0 | 0
  Life Threatening | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 56
Description: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Setmelanotide: PPL Group: Participants with POMC/PCSK1/LEPR biallelic mutations collectively referred as PPL received setmelanotide at a dose of 0.5 mg QD via SC injection for 52 weeks. The dose was escalated by increments of 0.5 mg every 2 weeks, if tolerated, at the dose escalation visits (Weeks 2, 4, and 6) to a maximum dose of 0.5 to 2.0 mg QD with the maximum dose based on body weight. Following the last dose in this study, participants who were considered likely to benefit from continued setmelanotide treatment and who had completed this trial could be eligible to enter an open-label long-term extension (LTE) trial with setmelanotide.
Arm/Group | Setmelanotide: PPL Group | Setmelanotide: BBS Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide: PPL Group (N=7) | Setmelanotide: BBS Group (N=5)
Nasopharyngitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 0
COVID-19 (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 2
Otitis media (Infections and infestations) | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1
Skin candida (Infections and infestations) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Injection site bruising (General disorders) | 1 | 3
Injection site pruritus (General disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 2
Injection site discoloration (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
Injection site erythema (General disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04966741/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04966741/SAP_001.pdf